CLINICAL TRIAL: NCT02660021
Title: Prospective Registry of 3-dimensional Virtual Treatment Planning of Orthognathic Surgery
Acronym: 3D-VIRTOG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Gwen Swennen, maxillofacial surgeon, MD, LDS, DMD, PhD, FEBOMFS, AZ Sint-Jan AV
Other Study IDs: B049201627035
Record Dates: First submitted 2016-01-11; First posted 2016-01-21 (Estimated); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Jaw Abnormalities
Keywords: three-dimensional virtual treatment planning; orthognathic surgery
MeSH Terms: conditions — Jaw Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
Orthognathic surgery or corrective jaw surgery is indicated for conditions of the jaw and face that are related to structure or growth malfunctioning, orthodontic problems, or co-morbidities associated with skeletal disfigurement.

Imaging is crucial in the assessment and treatment planning of orthognathic surgery patients. Until recently, two-dimensional (2D) imaging, through cephalometry, was standard practice. However, it showed several limitations. The introduction of the cone-beam computed tomography (CBCT) enabling three-dimensional (3D) imaging has caused a paradigm shift. Though widespread implementation in routine practice is not yet present. Our department is one of the pioneers in the world of 3D virtual treatment planning for orthognathic surgery. The "triple CBCT scan procedure" has been developed in-house and implemented already in 2009.

The investigators aim to develop a prospective database registering 3D treatment planning data of all consecutive patients eligible for orthognathic surgery, performed by Prof. Swennen. Patient demographics, detailed virtual 3D treatment planning parameters and orthognathic surgery data are being collected during consecutive visits within the framework of routine practice.

Development of a database registering 3D virtual treatment planning data of orthognathic surgery, will provide more information about potential patient, virtual planning and surgical factors influencing postoperative accuracy of jaw correction, long-term stability of the jawbone, long-term condylar resorption, or soft tissue response. In general, it could provide answers on research questions that have been examined in prior studies on 2D-imaging, but can now be re-examined in case of 3D-imaging. Moreover, registration of those results could function as a measurement of quality of care, or could be used for sample size calculation for future large multicenter prospective trials.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all ages
* Both female and male patients
* Patients should present themselves at the Department of Oral and Maxillofacial Surgery of the General Hospital Saint-John Bruges for orthognathic surgical treatment
* Patients receive standardized cone-beam computed tomography (CBCT) image acquisition (i-CAT, Imaging sciences international, inc, Hatfield, USA) according to the "triple" CBCT scan protocol
* Patients' orthognathic surgery should be prepared by a standardized setup of an augmented 3D virtual patient model in centric relation, with detailed occlusal and intercuspidation data using the "triple" voxel-based rigid registration protocol (Maxilim v2.2.2., Nobel Biocare c/o Medicim nv, Mechelen, Belgium)
* Patients' surgery should be prepared preoperatively through 3D virtual planning steps performed with the same software, by the same surgeon (GS)
* Patients should be operated by the same surgeon (GS)

Exclusion Criteria:

* All patients that do not fit in the abovementioned description
* Patients with posttraumatic deformity
* Patients with congenital deformity
* Patients with preprosthetic indication

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consenting patients, eligible for orthognathic surgery, performed at the General Hospital Saint-John Bruges, from July 1st 2010 onwards.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2010-07; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy of hard tissue, soft tissue and teeth transfer after 3D planning, as measured with CBCT | within 12 months postoperative

SECONDARY OUTCOMES:
Prevalence of patients with an indication for orthognathic surgery | 6 years
Accuracy of bone transfer, as measured through superimposition of 3D planning CBCT and postoperative CBCT | 4 weeks postoperative
Long-term stability, through clinical evaluation and superimposition of 3D planning CBCT and postoperative CBCT | 6 months postoperative
number of patients with condylar resorption | until 12 months postoperative
number of patients with temporomandibular joint complications | until 12 months postoperative

OTHER OUTCOMES:
sample size calculation for future large prospective trials, based on pilot data | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Gwen Swennen, MD, LDS, DMD, PhD, FEBOMFS, Principal Investigator — Maxillofacial Surgeon
Locations (1):
- General Hospital Saint-John Bruges, Bruges, Belgium

IPD SHARING:
Plan to Share IPD: No